CLINICAL TRIAL: NCT07067515
Title: Effectiveness of Omega-3 Poly Unsaturated Fatty Acids on The Treatment of Gingival Hyperpigmentation: A Randomized Controlled Clinical Trial
Brief Title: Effectiveness of Omega-3 Poly Unsaturated Fatty Acids on The Treatment of Gingival Hyperpigmentation
Acronym: Omega-3
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Suez Canal University; self funded (Other: no organization)
Record Dates: First submitted 2025-06-02; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Hyperpigmentation; Gingival Hyperpigmentaion
Keywords: depigmentation; omega 3; poly unsaturated fatty acids; racial pigmentation
MeSH Terms: conditions — Hyperpigmentation; Vitiligo | interventions — Fatty Acids, Unsaturated; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- surgical treatment (Active Comparator): Patients with gingival hyperpigmentation of oral mucosa. For the scalpel technique, following the administration of a local anesthetic solution, a partial split thickness flap was raised with the help of blade no. 15 with the Bard Parker handle to scrape the epithelium in maxillary anterior area from canine to canine in the other side; will be surgical removal of pigmentation using the scalpel in 45 degrees to remove the superficial layer. Bleeding Will be controlled using a pressure pack with sterile gauze. Care was taken that excessive tissue was not removed thereby avoiding any bone exposure. This will be followed by careful examination of the exposed connective tissue surface, and the wound will be irrigated with saline. Bleeding will be controlled using a pressure pack, and once hemostasis is achieved, the site will be covered by a periodontal dressing for a period of one week. patients will be advised to stop eating hard, acidic, spicy, and colored foods before surgery-
  Interventions: Procedure: surgical treatment
- non surgical with PUFA injection (Experimental): The hyperpigmented gingiva in the canine/1st premolar region to the contralateral comparable tooth region in the maxillary aesthetic areas will be the target area for this procedure. A local anesthesia will be used to numb the area. Using an insulin and plastic syringe (needle: 30-gauge, 8 mm length), 1-2 gram /0.1-0.2 ml of Omega-3 (PUFAs) will be injected into the gingiva at approximately the epithelial connective tissue interface until the tissue blanche, 2-3 mm apart. The insulin syringe, bevel facing upward, will be inserted into the corresponding gingival tissues. For four weeks, this dosage of omega-3 (PUFAs) will be administered once a week. Furthermore, patients will take 2 capsules. Each capsule contains 1 gram of Omega3(PUFAs) as an additional food supplement (up to 3 gram daily for the period of injection except the day of injection. the patients will receive a packet containing required number of capsules have to be taken every week.
  Interventions: Combination Product: non surgical with PUFA injection

INTERVENTIONS:
Combination Product: non surgical with PUFA injection — The hyperpigmented gingiva in the canine/1st premolar region to the contralateral comparable tooth region in the maxillary aesthetic areas will be the target area for this procedure. A local anesthesia will be used to numb the area. Using an insulin and plastic syringe (needle: 30-gauge, 8 mm length), 1-2 gram /0.1-0.2 ml of Omega-3 (PUFAs) will be injected into the gingiva at approximately the epithelial connective tissue interface until the tissue blanche, 2-3 mm apart. The insulin syringe, bevel facing upward, will be inserted into the corresponding gingival tissues. For four weeks, this dosage of omega-3 (PUFAs) will be administered once a week. Furthermore, patients will take 2 capsules. Each capsule contains 1 gram of Omega3(PUFAs) as an additional food supplement (up to 3 gram daily for the period of injection except the day of injection. the patients will receive a packet containing required number of capsules have to be taken every week.
  Arms: non surgical with PUFA injection
Procedure: surgical treatment — Patients with gingival hyperpigmentation of oral mucosa. For the scalpel technique, following the administration of a local anesthetic solution, a partial split thickness flap was raised with the help of blade no. 15 with the Bard Parker handle to scrape the epithelium in maxillary anterior area from canine to canine in the other side; will be surgical removal of pigmentation using the scalpel in 45 degrees to remove the superficial layer. Bleeding Will be controlled using a pressure pack with sterile gauze. Care was taken that excessive tissue was not removed thereby avoiding any bone exposure. This will be followed by careful examination of the exposed connective tissue surface, and the wound will be irrigated with saline. Bleeding will be controlled using a pressure pack, and once hemostasis is achieved, the site will be covered by a periodontal dressing for a period of one week. patients will be advised to stop eating hard, acidic, spicy, and colored foods before surgery. All patie
  Arms: surgical treatment

SUMMARY:
This new study compares the effectiveness of scalpel surgery and omega-3 poly unsaturated fatty acid (PUF) injections in treating gingival hyperpigmentation.

DETAILED DESCRIPTION:
Thirty patients complaining from gingival hyperpigmentation will be involved in this study. 30 patients will be divided into two groups each group will be randomly allocated into: Group(I) will be treated with intra-gingival tissue injection of 1-2grams of Omega-3 (PUFAs) every week. In addition to administering a daily dosage of two gram of Omega-3 (PUF) both prior to and following surgery. The second group (II) will be treated with surgical conventional technique to remove hyperpigmentation. Patients with mild to moderate hyperpigmented gingiva who are selected with maxillary esthetic area. Hyperpigmentation will be followed up at baseline, one month, 3 months and six months.

ELIGIBILITY:
Inclusion Criteria:

* Patients complained of mild to moderate gingival hyperpigmentation in the anterior area of maxilla.

.Systemically healthy subjects with Dummett and Bolden index score 1,2 and 3 having well-maintained oral hygiene, with aesthetic concern and willing to undergo minor surgical procedures.

* Adequate oral hygiene conditions.
* Age from 21-50 years old.
* All patients will be physically healthy with no medical history of any systemic disease that will contraindicate the use of omega-3 (PUFAs) or may complicate the healing process.
* Co-operative motivated patients

Exclusion Criteria:

* The patient with the following criteria will be excluded from the study:

  * patients complaining of sever gingival hyperpigmentation in the anterior area of maxilla.
  * Smokers.
  * Pregnant, lactating (breast feeding) women's.
  * Patient with allergy to anesthesia
  * Patients undergoing chemotherapy or radiotherapy

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-08-07 (Estimated); Study Completion 2025-08-28 (Estimated)

PRIMARY OUTCOMES:
Change in gingival pigmentation | measured at baseline, 1 month, 3 month and 6 months postoperative
  decrease melanin color of the gingiva and transform into regular pink color either by surgical; or non-surgical technique measured by The Dummett oral pigmentation (DOPI) (Dummett, 1945) for the intensity of oral pigmentation The scoring criteria as 0=Gingiva in pink color,1=Mild light brown gingival color,2=Medium gingival color or mixed (brown &pink) gingival color and 3=Deep brown /blue-black gingival color

SECONDARY OUTCOMES:
post operative pain | After the procedures, a day of procedures and a week of procedures
  measure the post operative pain at 10-point Visual Analogue Scale (VAS). from '0=No pain' to increasing pain intensity at '10=Worst pain
changes in gingival pigmentation distribution | base line ,1month,3 months and 6 months
  measure the changes in gingival pigmentation distribution by Hedin melanin index (Hedin, 1977) scoring criteria 0=No pigmentation,1=One or two solitary units,2=More than three units of pigmentation in the papillary gingiva without formation of a continuous ribbon,3=One or more short continuous ribbons of pigmentation and 4=One continuous ribbon including the entire area between the canines an interdental papilla with half of the marginal gingiva on either side
Gingival bleeding | At the time of procedures
  severity of gingival bleeding as assessed by the scoring criteria as follows: 0=No bleeding, 1=Isolated bleeding, 2=Mild bleeding, 3=Moderate or severe bleeding
wound healing | After a day of procedures and after a 7-10 day of procedures
  measure the post-operative wound healing are estimated and scored as follow :0= presence of necrotic gingival tissue ,1=presence of the ulcer in the gingiva, 2=incomplete gingival epithelization ,3=complete gingival epithelization

CONTACTS AND LOCATIONS:
Overall Officials: Assistant Professor of Oral Medicine and Periodontology, Principal Investigator — Suez Canal University; Lecturer of Oral medicine and Periodontology, Study Director — Suez Canal University
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Balcos, M.C., Kim, S.Y., Jeong, H.S., Yun, H.Y., Baek, K.J., Kwon, N.S., Park, K.C. and Kim, D.S., 2014. Docosahexaenoic acid inhibits melanin synthesis in murine melanoma cells in vitro through increasing tyrosinase degradation. Acta Pharmacologica Sini — https://www.bing.com/ck/a?!&&p=b33d114f981f97fc13862467968ac502c5149a84fe73c582cc521217a761ec04JmltdHM9MTc0NDU4ODgwMA&ptn=3&ver=2&hsh=4&fclid=0ecbbb60-da4a-6df3-1656-aa91db366c5e&psq=pubmed+search&u=a1aHR0cHM6Ly9wdWJtZWQubmNiaS5ubG0ubmloLmdvdi8&ntb=1
- Available data/document: Free PMC article. — https://pubmed.ncbi.nlm.nih.gov/31353554/
- Available data/document: PMC article. — https://pubmed.ncbi.nlm.nih.gov/30734608/
- Available data/document: Free PMC article. — https://pubmed.ncbi.nlm.nih.gov/35508275/